CLINICAL TRIAL: NCT00259116
Title: A Pilot Safety and Dose-Finding Trial of Intravenous Recombinant Human Relaxin (rhRlx) in Compensated Congestive Heart Failure
Brief Title: A Pilot Study of Recombinant Human Relaxin (rhRlx) in Compensated Congestive Heart Failure
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Corthera, Inc.(formerly BAS Medical, Inc.), a member of the Novartis group of companies (Industry)
Responsible Party: Sam Teichman, Chief Medical Officer, BAS Medical
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RLX.CHF.001
Record Dates: First submitted 2005-11-28; First posted 2005-11-29 (Estimated); Last update posted 2009-04-15 (Estimated); Status verified 2009-04

CONDITIONS: Heart Failure, Congestive
Keywords: Congestive heart failure; Relaxin; Cardiac hemodynamics
MeSH Terms: conditions — Heart Failure | interventions — Relaxin

INTERVENTIONS:
Drug: Relaxin

SUMMARY:
This trial is a single center, open-label, dose-finding study of recombinant human relaxin (rhRlx) given intravenously (IV) to patients with stable, compensated CHF.

DETAILED DESCRIPTION:
Serial cohorts of patients with stable CHF will be enrolled upon meeting eligibility criteria. Dose escalation will be guided by hemodynamic response, safety and tolerability. The effects of rhRlx on hemodynamics will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients over the age of 18
* New York Heart Association (NYHA) Class II-III CHF
* Left Ventricular Ejection Fraction (LVEF) of < 35%

Exclusion Criteria:

* Acute coronary syndrome
* Acute decompensated CHF
* Hypotension
* Recent significant arrhythmia
* Recent stroke
* Significant renal or hepatic impairment
* Pregnancy or child-bearing potential

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18
Dates: Start 2005-11

PRIMARY OUTCOMES:
Cardiac hemodynamics including PCWP, CO/CI, SVR

SECONDARY OUTCOMES:
Safety and tolerability
Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Sam Teichman, MD, Study Director — BAS Medical - Sponsor
Locations (1):
- Charite Hospital, Berlin, Germany